CLINICAL TRIAL: NCT07084233
Title: Effects of Mindfulness and Self-regulation Training on Anxiety, Depression, PTSD, and Leadership: a Randomized Controlled Trial in Ukraine
Brief Title: Effects of Mindfulness and Self-regulation Training on Anxiety, Depression, PTSD, and Leadership
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Ukrainian Catholic University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009491
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Depression Disorder; PTSD - Post Traumatic Stress Disorder
Keywords: anxiety; depression; post-traumatic stress disorder; sleep quality; self-regulation; mindfulness; trauma-informed; resilience
MeSH Terms: conditions — Anxiety Disorders; Combat Disorders; Depression; Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Self-Control

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMFT arm (Experimental): This arm will begin the three-week Mindfulness Mind Fitness Training course shortly after enrolling. This course consists of 7.5 hours of live, online, group instruction.
  Interventions: Behavioral: Mindfulness based, trauma informed, self-regulation skills training
- Waitlist-control (No Intervention): This arm will receive no intervention of any kind during the study. Once the study is complete, they will be able to enroll in the same MMFT course that the intervention arm received.

INTERVENTIONS:
Behavioral: Mindfulness based, trauma informed, self-regulation skills training — The study intervention, MMFT, consists of 7.5 hours of live, online courses, in three sessions, over three weeks. The entire intervention group (n=100) will participate in each session simultaneously, with four trainers and two translators.
  Session 1 (3 hours): This session will introduce three mind fitness exercises. Session 2 (3 hours): This session will begin with mind fitness practice and discussion about participants' experience with the exercises during the previous two weeks.
  Session 3 (1.5 hours): This session is for participants to integrate course content at an experiential level-no new content will be offered. The session will include some guided practice, but mostly focus on answering questions from participants and/or providing guidance to participants for how to navigate challenges with practice.
  During the three weeks participants are in the course, they will be asked to practice the MMFT techniques for 5-60 minutes per day.
  Arms: MMFT arm

SUMMARY:
The goal of this study is to measure the effects of Mindfulness-based Mind Fitness Training (MMFT) on anxiety, depression, post-traumatic stress disorder, sleep quality, and leadership.

DETAILED DESCRIPTION:
Globally, depressive disorders were the second highest cause of years lost to disability in 2021, having increased 36.5% since 2010, and anxiety disorders were sixth. Furthermore, 4% of the global population has had post-traumatic stress disorder at some point in their lives. In conflict-affected settings, such as Ukraine, the prevalence of these disorders can be especially high: 47% depression, 54% anxiety, and over 50% PTSD. Given this high mental illness burden, widespread disruption caused by Russian attacks, and a historically under-resourced mental health care system. Ukraine is an ideal setting to test novel digital mental health interventions (DMHIs) that can be delivered either standalone or by non-clinicians, and that may hold potential for other populations stressed and traumatized by armed conflict, natural disasters, and displacement.

Recent meta-analyses show that DMHIs reduce symptomology associated with anxiety disorders, depression, and PTSD. However, effects vary as a result of several factors, including populations targeted, level of support provided, and technology used. Furthermore, investigation of underlying mechanisms has mostly examined internet-based cognitive behavioral therapy, leaving the mechanisms active in other therapeutic approaches poorly understood.

The investigators propose to test a DMHI called Mindfulness-based Mind Fitness Training (MMFT) in the Ukrainian context. MMFT was designed with two goals in mind: (1) to improve self-regulation and resilience by widening individuals' windows of tolerance to stress arousal; and (2) to do so in a trauma/dysregulation-informed manner. MMFT cultivates two core skills, attentional control and tolerance for challenging experience, through (1) an understanding of the neurobiology of stress, trauma, and resilience; (2) mindfulness skills training; (3) body-based self-regulation skills training, drawn from body-based trauma therapies such as sensorimotor psychotherapy and Somatic Experiencing; and (4) concrete applications for daily life. MMFT's body-based self-regulation exercises, as well as its unique exercise sequence to gradually cultivate interoceptive awareness, make it distinct from other mindfulness-based interventions. This focus on grounding and gradual cultivation of interoceptive awareness is particularly important for populations with significant prior exposure to prolonged or overwhelming stress, so that they do not inadvertently become re-traumatized. A small pilot in early 2024, suggests MMFT is applicable and feasible in wartime Ukraine.

The investigators will randomize 200 participants in a 1:1 ratio to (i) a three-week MMFT course, or (ii) a waitlisted control group. Immediately prior to the course, all participants will complete a baseline questionnaire on demographics, anxiety, depression, post-traumatic stress disorder, sleep quality, and leadership. Three weeks later, after group (i) has completed the course, both groups will complete a similar endline questionnaire. Intention-to-treat analysis will be used to test for an effect of MMFT on anxiety, depression, post-traumatic stress disorder, sleep quality, and leadership.

The secondary objective of the study is to qualitatively understand participant experience of the sessions and of the three MMFT exercises, including their attitudes towards these sessions and their experience of the impacts. A small subset of the MMFT group (~10 participants) will be randomly selected to take part in a one-time in-depth interview, lasting 30-60 minutes. Interview content will cover participant experience with the intervention, their reaction to the content and to the MMFT trainers, discussion of any barriers or challenges that they faced, and descriptions of any changes that they notice.

ELIGIBILITY:
Inclusion Criteria:

* Ukrainian speaker resident in Ukraine

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Depression | T1 (time of enrollment) [i.e. immediately prior to randomization]; T2 (three weeks post-randomization) [i.e. immediately post completion of intervention in the intervention group]
  Change in PHQ-9 (Patient Health Questionnaire-9) over three weeks. This 9-item self-report scale asks how often, over the past two weeks, respondents experienced core depressive symptoms; each item is rated 0-3 ("Not at all" to "Nearly every day") and summed for a total severity score ranging from 0 to 27.
Post-traumatic stress disorder symptoms | T1 (time of enrollment) [i.e. immediately prior to randomization]; T2 (three weeks post-randomization) [i.e. immediately post completion of intervention in the intervention group]
  Change in post-traumatic stress over three weeks. The PCL-5 self-report measure uses a Likert scale (0-4) to quantify the extent to which the respondent is bothered by 20 PTSD-related symptoms that are summed for a total severity score of 0 to 80.
Anxiety | T1 (time of enrollment) [i.e. immediately prior to randomization]; T2 (three weeks post-randomization) [i.e. immediately post completion of intervention in the intervention group]
  Change in GAD-7 (Generalized Anxiety Disorder-7) over three weeks. This 7-item self-report measure uses the same 0-3 Likert scale to capture the frequency of common anxiety symptoms in the past two weeks, yielding a total score of 0 to 21 that reflects overall anxiety severity.

SECONDARY OUTCOMES:
Sleep quality | T1 (time of enrollment) [i.e. immediately prior to randomization]; T2 (three weeks post-randomization) [i.e. immediately post completion of intervention in the intervention group]
  Change in Pittsburgh Sleep Quality Index (PSQI) over three weeks. This self-report instrument assesses sleep quality over the past month by combining 19 items into seven component scores (e.g., latency, duration, disturbances), each rated 0-3; the components are summed for a global score of 0 to 21, with higher totals indicating poorer overall sleep quality.
Leadership character | T1 (time of enrollment) [i.e. immediately prior to randomization]; T2 (three weeks post-randomization) [i.e. immediately post completion of intervention in the intervention group]
  Change in character dimensions of leadership over three weeks. Participants self-report how frequently they apply each of eleven dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ukrainian Catholic University, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plessen CY, Panagiotopoulou OM, Tong L, Cuijpers P, Karyotaki E. Digital mental health interventions for the treatment of depression: A multiverse meta-analysis. J Affect Disord. 2025 Jan 15;369:1031-1044. doi: 10.1016/j.jad.2024.10.018. Epub 2024 Oct 15. PMID 39419189
- [Background] Stanley, EA. (2019). Widen the Window: Training Your Brain and Body to Thrive during Stress and Recover from Trauma. Avery Books.